CLINICAL TRIAL: NCT07227337
Title: Being Safe, Healthy, And Positively Empowered (BSHAPE): A Digital Multicomponent Intervention to Improve Health and Safety Outcomes Among Women With Cumulative Exposures to Violence
Brief Title: Being Safe, Healthy, And Positively Empowered (BSHAPE) Intervention Study
Acronym: BSHAPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00504423; 1R01MD018503-01A1 (NIH)
Record Dates: First submitted 2025-11-10; First posted 2025-11-12 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Post Traumatic Stress Disorder; Depression; Violence
Keywords: Post Traumatic Stress Disorder (PTSD); Depression; Violence
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): Participants will be randomized to the Control Arm
  Interventions: Other: Control (general wellness)
- BSHAPE intervention (Experimental): Participants will be randomized to the BSHAPE intervention.
  Interventions: Behavioral: BSHAPE

INTERVENTIONS:
Behavioral: BSHAPE — BSHAPE is designed to comprehensively assess cumulative exposures to violence, evaluate current safety needs, and provide components to mitigate trauma-related symptoms (e.g., mental health challenges, HIV/STI risk). It promotes health and resilience through psycho-education, skill-building, and mindfulness-based stress reduction practices.
  Arms: BSHAPE intervention
Other: Control (general wellness) — The control group will receive nutrition information and exercise guidance as well as a standard list of community resources.
  Arms: Control Arm

SUMMARY:
The purpose of the study is to evaluate a trauma informed digital multicomponent intervention design to improve health and safety outcomes for women with lifetime exposures to violence and co-occurring PTSD and/or depression symptoms

DETAILED DESCRIPTION:
Individuals with cumulative exposures to interpersonal violence are at high risk for co-occurring mental and physical health problems (e.g., PTSD, HIV/STI) and safety issues such as living in unsafe households or being in unsafe relationships. The proposed research will test the efficacy of Being Safe, Healthy, and Positively Empowered (BSHAPE), an intervention designed to comprehensively assess cumulative exposures to violence, current safety needs, and includes components to reduce the impact of trauma such as poor mental health, HIV/STI risk, and to promote health through knowledge building, skill building, and stress reduction practices.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* foreign-born immigrant woman
* self-reported history of cumulative exposure to violence, and presence of PTSD and/or depression symptoms

Exclusion Criteria:

* Participants who don't meet the above criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender women
Enrollment: 676 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress as Assessed by The Perceived Stress Scale-10 (PSS-10) | Baseline (1st month), 3, 6 and 12 months
  The Perceived Stress Scale-10 (PSS-10) is a 10-item questionnaire that measures the degree to which situations in one's life are appraised as stressful. Total scores range from 0 to 40, with higher scores indicating higher levels of perceived stress.
Depression as Assessed by The Patient Health Questionnaire-9 (PHQ-9) | Baseline (1st month), 3, 6 and 12 months
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item self-report questionnaire that measures depression severity over the past 2 weeks. Total scores range from 0 to 27, with higher scores indicating more severe depression symptoms. Scores can be categorized as: minimal depression (0-4), mild depression (5-9), moderate depression (10-14), moderately severe depression (15-19), or severe depression (20-27).
PTSD as Assessed by The PTSD Checklist-Civilian Version (PCL-C) | Baseline (1st month), 3, 6 and 12 months
  The PTSD Checklist-Civilian Version (PCL-C) is a 17-item self-report questionnaire that measures provisional PTSD over the past month. Total scores range from 17 to 85, with higher scores indicating greater PTSD symptom severity.
Self-Protection Behavior Checklist | Baseline (1st month), 3, 6 and 12 months
  The Self-Protection Behavior Checklist is a 6-item self-report questionnaire that measures the frequency of self-protective strategies used by participants. Total scores range from 0 to 24, with higher scores is better, indicating more frequent use of self-protective strategies.
Empowerment for Safety as Assessed by The Adapted Measure of Victim Empowerment Related to Safety (MOVERS) | Baseline (1st month), 3, 6 and 12 months
  The Measure of Victim Empowerment Related to Safety (MOVERS) is a 12-item self-report questionnaire that measures survivor empowerment within the domain of safety. Total scores range from 12 to 60, with higher scores indicating greater empowerment for safety.
Self-Care Behaviors as Assessed by The Mindful Self-Care Scale (MSCS) and The Behavioral Activation for Depression Scale-Short Form (BADS-SF) | Baseline (1st month), 3, 6 and 12 months
  The Self-Care Behaviors Scale is a 23-item self-report measure assessing engagement in self-care behaviors across multiple domains, including mindful relaxation, supportive relationships, supportive structure, general, and clinical areas. The scale combines items from the Mindful Self-Care Scale (MSCS) and the Behavioral Activation for Depression Scale-Short Form (BADS-SF) into a single composite measure. Total scores are calculated as the sum of all items and range from 0-92, with higher scores indicating greater engagement in self-care behaviors.

SECONDARY OUTCOMES:
Safe Sex Behavior as Assessed by The Safe Sex Behavior Questionnaire (SSBQ) | Baseline (1st month), 3, 6 and 12 months
  The Safe Sex Behavior Questionnaire (SSBQ) is a 24-item self-report questionnaire that measures sexual behaviors, condom usage, high risk sexual behaviors, and sexual communication and negotiation. Total scores range from 24 to 96, with higher scores indicating greater frequency of use of safe sex practices.
Cognitive and Affective Mindfulness as Assessed by The Adapted Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) | Baseline (1st month), 3, 6 and 12 months
  The Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) is a 12-item self-report questionnaire that measures individual differences in mindfulness. Total scores range from 12 to 48, with higher scores indicating greater mindfulness abilities.
Resilience as Assessed by The Brief Trauma Resiliency Scale (BTRS) | Baseline (1st month), 3, 6 and 12 months
  The Brief Trauma Resiliency Scale (BTRS) is a 28-item self-report questionnaire that measures trauma resilience, ability to "bounce back," after a traumatic experience. Total scores range from 28 to 140, with higher scores indicating greater trauma resilience.
Health-related Self-Care Efficacy as Assessed by The Self-Care Self-Efficacy Scale (SCSES) | Baseline (1st month), 3, 6 and 12 months
  The Self-Care Self-Efficacy Scale (SCSES) is a 10-item self-report questionnaire that measures individuals' confidence in their ability to engage in self-care behaviors across various health contexts. Total scores range from 10 to 50, with higher scores indicating greater confidence in performing self-care behaviors.
Trauma Coping Self-Efficacy as Assessed by Trauma Coping Self-Efficacy (CSE-T) | Baseline (1st month), 3, 6 and 12 months
  The Trauma Coping Self-Efficacy Scale is a 9-item self-report questionnaire that measures an individual's perceived confidence in their ability to cope with and recover from traumatic experiences. Total scores range from 9 to 63, with higher scores indicating greater confidence in one's ability to cope with trauma-related challenges and engage in recovery processes.
General Self-Efficacy as Assessed by The General Self-Efficacy Scale-Short Form (GSE-6) | Baseline (1st month), 3, 6 and 12 months
  The General Self-Efficacy Scale-Short Form (GSE-6) is a 6-item self-report questionnaire. The scale assesses a general sense of perceived self-efficacy with the aim in mind to predict coping with daily hassles as well as adaptation after experiencing all kinds of stressful life events. Total scores range from 6 to 24, with higher scores indicating greater general self-efficacy beliefs
Emotion Regulation as Assessed by The Emotion Regulation Questionnaire (ERQ) | Baseline (1st month), 3, 6 and 12 months
  The Emotion Regulation Questionnaire (ERQ) is a 10-item self-report questionnaire that measures individual differences in emotion regulation strategies. Total scores range from 10 to 70, with higher scores indicating greater overall use of emotion regulation strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Bushra Sabri, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No